CLINICAL TRIAL: NCT03692234
Title: Homoarginine in Stroke (HiS) Study
Brief Title: Homoarginine Supplementation in Patients After Stroke
Acronym: HiS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Homoarginine in Stroke
Record Dates: First submitted 2018-07-18; First posted 2018-10-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Deficiency; Diet
Keywords: homoarginine
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: randomized double-blind placebo controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo capsules containing lactose - oral once weekly administration for six month
  Interventions: Other: placebo
- homoarginine (Active Comparator): 125 mg L-homoarginine supplement - oral once weekly administration for six month
  Interventions: Dietary Supplement: 125 mg L-homoarginine

INTERVENTIONS:
Dietary Supplement: 125 mg L-homoarginine — capsules for oral supplementation
  Arms: homoarginine
Other: placebo — capsules for oral supplementation
  Arms: placebo

SUMMARY:
This study represents a follow-up of the previous study "Single and Multiple Doses of an Oral Formulation of L-Homoarginine in Healthy Human Subjects" (NCT02675660). This study will evaluate the applicability of an oral formulation of L-homoarginine to normalize homoarginine blood levels in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke (CT or MRI), high-risk transient ischemic attack (ABCD2-score >= 4) or acute central retinal artery occlusion
* serum homoarginine </= 2.1 umol/L
* signed informed consent

Exclusion Criteria:

* no acute stroke
* serum homoarginine > 2.1 umol/L
* heart failure (NYHA > 1)
* chronic kidney disease (GFR <60 mL/min)
* not competent
* pregnancy, lactation
* no or withdrawn signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Homoarginine serum concentration | six month
  Normalization of homoarginine serum concentration to levels >2.1 umol/L.

SECONDARY OUTCOMES:
Intima-media thickness | six month
  Intima-media thickness (IMT) measured at both common carotid arteries using an edge detection system. Plaques are defined as protrusion of ≥1.5 mm in common, internal and external carotid artery.
National Institute of Health Stroke Scale | six month
  National Institute of Health Stroke Scale (NIHSS) will be assessed by a neurologist. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 (normal) and 4 (maximum impairment). The maximum possible score is 42, with the minimum score being a 0.
Modified Ranking Scale | six month
  Modified Ranking Scale (mRS) is a scale for measuring the degree of disability of a stroke patients. The scale runs from 0 (perfect health) to 6 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atzler D, Schonhoff M, Cordts K, Ortland I, Hoppe J, Hummel FC, Gerloff C, Jaehde U, Jagodzinski A, Boger RH, Choe CU, Schwedhelm E. Oral supplementation with L-homoarginine in young volunteers. Br J Clin Pharmacol. 2016 Dec;82(6):1477-1485. doi: 10.1111/bcp.13068. Epub 2016 Sep 20. PMID 27434056